CLINICAL TRIAL: NCT01948440
Title: ASI-MV Solutions: A Tailored Program for Substance Abusers in Early Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Responsible Party: Principal Investigator, Emil Chiauzzi, Vice President of Product Strategy, Inflexxion, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2R44DA026232-02 (NIH)
Record Dates: First submitted 2010-07-27; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Substance Abuse Treatment for Adults
Keywords: Substance abuse, early recovery, relapse prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASI-MV Solutions (Experimental): The Experimental group will complete the ASI-MV and use the ASI-MV Solutions program for eight 30-minute sessions, followed by monthly booster sessions. The Experimental group will undergo a baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention.
  Interventions: Behavioral: ASI-MV Solutions
- Treatment as Usual (No Intervention): The Control group participants will complete the ASI-MV and receive their normal course of treatment. The Control group will undergo a baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention.

INTERVENTIONS:
Behavioral: ASI-MV Solutions — The Experimental group will complete the ASI-MV and use the ASI-MV Solutions program for eight 30-minute sessions, followed by monthly booster sessions. The Experimental group will undergo a baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention.
  Arms: ASI-MV Solutions

SUMMARY:
Making referrals to medical and psychosocial services for substance abuse clients has proven difficult due to lack of access to services, inadequate counselor knowledge, and lack of motivation and skills among clients. Inflexxion is proposing the development of ASI-MV Solutions, which will educate clients about employment, legal, psychiatric, relapse prevention, medical, and family issues, as well as include resources and strategies for counselors. By linking learning modules to client results on the ASI-MV, an online interactive version of the ASI administered in treatment settings, we will be able to offer clients important tools to address key recovery issues and encourage counselors to make appropriate referrals to medical and psychosocial services.

DETAILED DESCRIPTION:
Substance abuse research indicates that: (1) addressing medical and psychosocial problems associated with substance abuse and dependence leads to better outcomes; (2) treatments are now shorter due in part to rising healthcare costs, and it is difficult to address these issues effectively during treatment, making medical and psychosocial ("wraparound") services following treatment essential; (3) counselors may lack the knowledge to effectively integrate these services; and (4) referrals to these services have been underutilized and clients may lack the motivation, knowledge, or skills to follow up with the referrals when they are made. To address these deficits, we are proposing the development of ASI-MV Solutions, which will provide tailored motivational feedback and skill-building lessons to clients to address specific psychosocial and medical problem areas. We expect that ASI-MV Solutions will have seven modules (Alcohol, Drugs, Medical, Psychiatric, Legal, Employment, and Family) corresponding to domains of the ASI-MV, a Web-enabled interactive version of the ASI administered in treatment settings. Substance abusers who have high severity scores on ASI-MV subscales will be directed to corresponding interactive lessons and local resources on ASI-MV Solutions. To demonstrate the feasibility of the program concept, the Phase I study focused on the Employment domain. All feasibility criteria were met and findings indicated: (1) Proposed content was based on highly positive findings from concept mapping, as well as usability and acceptance testing with clients and experts. Ratings of potential effectiveness and appeal were high. (2) Usability testing indicated that the program was usable by the target audience, the skills and outcomes were relevant to the target audience, and the program was regarded as potentially very helpful to the treatment process. We surpassed feasibility benchmarks for both clients and experts. (3) Our technical/design team produced a demonstration program that was perceived by key stakeholders as highly usable and engaging multimedia program, as well as determining the necessary technologies to produce the complete program in Phase II. In Phase II we will develop ASI-MV Solutions content, complete the ASI-MV Solutions program, field test the program, and conduct satisfaction and acceptance testing of the program with clients and counselors.

ELIGIBILITY:
Inclusion Criteria:

* Client Inclusion Criteria. We will recruit participants in the same proportions as in usability testing - 40% female, 40% minorities. The inclusion criteria for clients are the same as those for usability testing, except that we will require the participant to provide: (1) the names of at least three contacts who can help locate the client during the study, and (2) multiple means of contacting them (telephone, mail, and/or email). As with usability participants, we will seek clients who are in the early stages of treatment (30 days or less, including new intakes).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
improved outcomes, as measured by substance use, psychosocial, and psychological functioning | baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention
  Addiction Severity Index - Multimedia Version (ASI-MV)
greater problem-services matching, as measured by the number and fit of referred/received services | baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention
  Treatment Services Checklist (Client Version) and Treatment Services Checklist (Counselor Version).
greater treatment motivation | baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention
  Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES, Version 8D; Miller & Tonigan, 1996)
greater self-efficacy in managing psychosocial issues | baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention
  Drug Avoidance Self-Efficacy Scale

SECONDARY OUTCOMES:
treatment compliance | baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention
  Treatment Compliance: We will ask counselors to record scheduled and planned sessions within the treatment facility as a way of assessing treatment compliance. We will also ask counselors to record client reasons for leaving treatment prematurely (Against Medical Advice, moving, hospitalization, etc.).
treatment alliance with counselors | baseline assessment and one-month post-baseline, two-month post-baseline, and six-month post-intervention
  Working Alliance Inventory-Short Form (Clients) and Working Alliance Inventory-Short Form (Counselors)

CONTACTS AND LOCATIONS:
Overall Officials: Emil Chiauzzi, PhD, Principal Investigator — Inflexxion, Inc.